CLINICAL TRIAL: NCT02583594
Title: A Phase 1, Exploratory, Randomized, Open-label, 2-Arm Study to Characterize the Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Alemtuzumab 12mg Administered Subcutaneously or Intravenously in Patients With Progressive Multiple Sclerosis
Brief Title: A Study to Characterize Subcutaneous or Intravenous Alemtuzumab in Patients With Progressive Multiple Sclerosis
Acronym: SCALA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDU14260; 2015-002550-12 (EudraCT Number); U1111-1171-7939 (Other: UTN)
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Acyclovir; Methylprednisolone; Acetaminophen; Loratadine; ceterizine hydrochloride; dexchlorpheniramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- alemtuzumab (subcutaneous injection) (Experimental): Dose 1 (initial course) of alemtuzumab will be administered subcutaneously on 5 consecutive days, followed by Dose 2 (second course) on 3 consecutive days administered 12 months after initial course. Pre-medications (methylprednisolone, antihistamine [loratadine, cetirizine, dexchlorpheniramine], paracetamol, acyclovir) will be administered prior alemtuzumab administration.
  Interventions: Drug: Acyclovir; Drug: Methylprednisolone; Drug: alemtuzumab GZ402673; Drug: Paracetamol; Drug: Loratadine; Drug: Ceterizine; Drug: Dexchlorpheniramine
- alemtuzumab (intravenous infusion) (Experimental): Dose 1 (initial course) of alemtuzumab will be administered intravenously on 5 consecutive days, followed by Dose 2 (second course) on 3 consecutive days administered 12 months after initial course. Pre-medications (methylprednisolone, antihistamine [loratadine, cetirizine, dexchlorpheniramine], paracetamol, acyclovir) will be administered prior alemtuzumab administration.
  Interventions: Drug: Acyclovir; Drug: Methylprednisolone; Drug: alemtuzumab GZ402673; Drug: Paracetamol; Drug: Loratadine; Drug: Ceterizine; Drug: Dexchlorpheniramine

INTERVENTIONS:
Drug: Acyclovir — Pharmaceutical form:tablet Route of administration: oral
Drug: Methylprednisolone — Pharmaceutical form:tablet Route of administration: oral
Drug: alemtuzumab GZ402673 — Pharmaceutical form:solution for infusion Route of administration: intravenous
  Arms: alemtuzumab (intravenous infusion)
Drug: alemtuzumab GZ402673 — Pharmaceutical form:injection Route of administration: subcutaneous
  Arms: alemtuzumab (subcutaneous injection)
Drug: Paracetamol — Pharmaceutical form:tablet Route of administration: oral
Drug: Loratadine — Pharmaceutical form:tablet Route of administration: oral
Drug: Ceterizine — Pharmaceutical form:tablet Route of administration: oral
Drug: Dexchlorpheniramine — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

* To characterize the pharmacodynamic profile of 2 treatment courses of alemtuzumab administered by subcutaneous injection and 2 treatment courses of alemtuzumab administered by intravenous infusion in patients with progressive multiple sclerosis.

Secondary Objectives:

* To characterize the pharmacokinetic profiles of alemtuzumab administered by subcutaneous injection or intravenous infusion to patients with progressive multiple sclerosis.
* To characterize the safety and tolerability of alemtuzumab administered by subcutaneous injection or intravenous infusion to patients with progressive multiple sclerosis.

DETAILED DESCRIPTION:
The duration of study per patient will be approximately 61 months.

ELIGIBILITY:
Inclusion criteria:

* Male or female adults with a diagnosis of Multiple Sclerosis (MS) based on 2010 revision of McDonald criteria.
* Diagnosis of progressive MS including primary progressive MS and secondary progressive MS.
* Age ≥18 years.
* Signed informed consent form.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision.

Exclusion criteria:

* Patients with relapsing remitting MS.
* Any prior treatment with alemtuzumab or other anti-CD52 antibodies.
* Treatment with natalizumab in the 4 months prior to Study Visit 1.
* Progressive multifocal leukoencephalopathy (PML), or any clinical or imaging signs possibly indicative of undiagnosed PML. Particular vigilance is needed for patients with prior natalizumab exposure, even if the last exposure was more than 4 months prior to Study Visit 1.
* Treatment with methotrexate, azathioprine, or cyclosporine in the past 6 months.
* Treatment with mitoxantrone, cyclophosphamide, cladribine, rituximab, or any other immunosuppressant or cytotoxic therapy (other than steroids) in the last 12 months, or determined by the treating physician to have residual immune suppression from these treatments.
* Treatment with glatiramer acetate or interferon beta in the past 4 weeks.
* Treatment with fingolimod within the past 2 months.
* Treatment with dimethyl fumarate in the past 4 weeks.
* Treatment with teriflunomide within the past 12 months unless the patient has completed an accelerated clearance with cholestyramine or activated charcoal.
* Any known contraindications to the symptomatic therapy used in the infusion management guidance for this study.
* Hypersensitivity or contraindication to acyclovir.
* History of a hypersensitivity reaction other than localized injection site reaction to any biological molecule.
* If female, pregnancy (defined as positive β-HCG blood test) or lactating or breast-feeding.
* Current participation in another investigational interventional study.
* Any significant change in chronic treatment medication (ie, new chronic medication) within 14 days before inclusion.
* An investigational medicinal product within 3 months or 5 half-lives, whichever is longer, before study inclusion.
* Total lymphocyte or CD3+ counts are below normal limits at screening. If abnormal cell count(s) return to within normal limits, eligibility may be reassessed.
* Live, attenuated vaccine within 3 months prior to the randomization (Day 1) visit, such as varicella-zoster, oral polio, rubella vaccines.
* Any clinically relevant findings in the physical examination, medical history, or laboratory assessments which would compromise the safety of the patient.
* Women of childbearing potential not protected by highly-effective method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Latent or active tuberculosis infection, verified by testing as per local practice.
* Infection with human immunodeficiency virus (HIV).
* Known Hepatitis B (HBV) or Hepatitis C (HCV) infection.
* Active infection, eg, deep tissue infection, that the Investigator considers sufficiently serious to preclude study participation.
* Prior history of invasive fungal infections.
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any patient in the exclusion period of a previous study according to applicable regulations.
* Any patient who cannot be contacted in case of emergency.
* Any patient who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12-06 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the CD3+ lymphocyte subset after alemtuzumab administration | Baseline, 30 days after each treatment course

SECONDARY OUTCOMES:
Change from baseline in lymphocyte subsets after alemtuzumab administration | Baseline, 30 days after each treatment course
Change from baseline in total lymphocyte count after alemtuzumab administration | Baseline, 30 days after each treatment course
Change from baseline in helper/suppressor ratio after alemtuzumab administration | Baseline, 30 days after each treatment course
Assessment of pharmacokinetic parameter after alemtuzumab administration: maximum plasma concentration observed (Cmax) | 30 days after each treatment course
Assessment of pharmacokinetic parameter after alemtuzumab administration: time to reach Cmax (Tmax) | 30 days after each treatment course
Assessment of pharmacokinetic parameter after alemtuzumab administration: area under plasma concentration versus time curve from time zero until the last measurable concentration (AUClast) | 30 days after each treatment course
Assessment of pharmacokinetic parameter after alemtuzumab administration: area under plasma concentration (AUC) | 30 days after each treatment course
Assessment of pharmacokinetic parameter after alemtuzumab administration: terminal half-life (t1/2z) | 30 days after each treatment course
Number of patients with adverse events | 4 years
Number of patients with adverse events of special interest | 4 years
Number of patients with injection site reactions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 724001, Barcelona, Spain

REFERENCES:
- [Derived] Montalban X, Rodriguez-Acevedo B, Nos C, Resina M, Forner M, Wu Y, Chirieac M. SCALA: a randomized phase I trial comparing subcutaneous and intravenous alemtuzumab in patients with progressive multiple sclerosis. Ther Adv Neurol Disord. 2024 Nov 6;17:17562864241291655. doi: 10.1177/17562864241291655. eCollection 2024. PMID 39513023